CLINICAL TRIAL: NCT05023252
Title: Passive Mobile Self-Tracking of Mental Health by Veterans With Serious Mental Illness
Brief Title: Mobile Self-Tracking of Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 19-392
Record Dates: First submitted 2021-08-16; First posted 2021-08-26 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia; Bipolar Disorder; Schizoaffective Disorder; Post-traumatic Stress Disorder
Keywords: Mental health care; Informatics; Predictive Modeling; Bipolar disorder; Psychotic Disorders; Machine learning
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants in the trial are enrolled in an intervention group for 9 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mobile application (Experimental): Participants use a mobile application on their smartphone
  Interventions: Other: mobile application

INTERVENTIONS:
Other: mobile application — VetThrive is a mobile smartphone application that monitors and transmits mobile sensor and utilization data. This app is deployed in Veteran patients who passively self-track their behaviors and psychiatric symptoms.
  Other Names: VetThrive

SUMMARY:
Serious mental illnesses require years of monitoring and adjustments in treatment. Stress, substance abuse or reduced medication adherence cause rapid worsening of symptoms, with consequences that include job loss, homelessness, suicide, incarceration, and hospitalization. Treatment visits can be infrequent. Illness exacerbations usually occur with no clinician awareness, leaving little opportunity to make treatment adjustments. Tools are needed that quickly detect illness worsening. At least two thirds of Veterans with serious mental illness use a smartphone. These phones generate data that characterize sociability, activity and sleep. Changes in these are warning signs for relapse. Members of this project developed an app that monitors and transmits these mobile data. This project studies passive mobile sensing that allows Veterans to self-track their activities, sociability and sleep; and studies whether this can be used to track symptoms. The project intends to produce a mobile platform that monitors the clinical status of patients, identifies risk for relapse, and allows early intervention.

DETAILED DESCRIPTION:
Background: Serious mental illnesses are common, disabling, challenging to treat, and require years of monitoring with adjustments in treatments. Stress or reduced medication adherence can lead to rapid worsening in symptoms and functioning with consequences that include relapse, job loss, homelessness, incarceration, hospitalization and suicide. In usual care, clinician visits are infrequent, with intervals ranging from monthly to yearly. Communication between patients and clinicians between visits is challenging and often nonexistent. Patient illness exacerbations and relapses generally occur with little or no clinician awareness in real time, leaving little opportunity to adjust treatments.

Significance/Impact: For the large population of Veterans with serious mental illness, tools are needed that passively monitor their mental health status, allowing them to self-track their behaviors, quickly detect worsening of mental health, and support prompt assessment and intervention. At least 60% of Veterans with serious mental illness use a smart phone. These generate data that characterize sociability, activity, and sleep. Changes in these behaviors are warning signs of relapse. Passive self-tracking could be used to identify and predict worsening of illness in real time.

Innovation: Passive mobile sensing is a novel approach to illness self-tracking and monitoring. There has been relatively little research on passive self-tracking in serious mental illness, with limited analytics development in this area, and none in VA.

Specific Aims: This project studies passive mobile sensing with Veterans in treatment for serious mental illness. Data are used for self-tracking of behaviors and symptoms. While passive mobile sensing has been feasible, acceptable and safe in patients with serious mental illness, these are studied for the first time in VA. Analytics are developed that use passive data to predict behaviors and symptoms. This project responds to the HSR&D priority areas of Mental Health and Healthcare Informatics. The project has these objectives:

1. Conduct user-centered design of passive mobile self-tracking to support Veterans' management of their mental health.
2. Study the feasibility, acceptability and safety of passive self-tracking of mental health that includes feedback of mental health status to the Veteran.
3. Use mobile sensor and phone utilization data to develop individualized estimates of sociability, activities, and sleep as measured by weekly interviews.
4. Study the predictive value of using data on sociability, activities, and sleep to identify exacerbations of psychiatric symptoms.

Methodology: Activities can be assessed with data on movement, location, and habits. Sociability can be assessed with data on communication and public interactions. Sleep can be assessed using data on light, sound, movement, and phone use. Investigators on this project developed a functional mobile app that monitors and transmits mobile sensor and utilization data. Focus groups and in-lab usability testing inform further app and intervention development. Mixed methods research study deployment in Veterans who passively self-track their behaviors and psychiatric symptoms. If this project meets intended goals, the VA will have a mobile analytics platform that continuously monitors behaviors and symptoms of patients with serious mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Veteran patient at the Greater Los Angeles Veterans Healthcare Center with a chart diagnosis of serious mental illness, defined as a diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder
* Risk for symptoms based on having had, during the past year, psychiatric hospitalization, psychiatric emergency care, lived at a crisis program, or more than 6 outpatient visits; and,
* Ownership of a smartphone with a data plan

Exclusion Criteria:

* Under age 18
* Has a conservator/legally authorized representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stehle Young, MD MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Young AS, Choi A, Cannedy S, Hoffmann L, Levine L, Liang LJ, Medich M, Oberman R, Olmos-Ochoa TT. Passive Mobile Self-tracking of Mental Health by Veterans With Serious Mental Illness: Protocol for a User-Centered Design and Prospective Cohort Study. JMIR Res Protoc. 2022 Aug 5;11(8):e39010. doi: 10.2196/39010. PMID 35930336
- [Result] Medich M, Cannedy SL, Hoffmann LC, Chinchilla MY, Pila JM, Chassman SA, Calderon RA, Young AS. Clinician and Patient Perspectives on the Use of Passive Mobile Monitoring and Self-Tracking for Patients With Serious Mental Illness: User-Centered Approach. JMIR Hum Factors. 2023 Oct 24;10:e46909. doi: 10.2196/46909. PMID 37874639
- [Result] Lin Z, Weinberger E, Nori-Sarma A, Chinchilla M, Wellenius GA, Jay J. Daily heat and mortality among people experiencing homelessness in 2 urban US counties, 2015-2022. Am J Epidemiol. 2024 Nov 4;193(11):1576-1582. doi: 10.1093/aje/kwae084. PMID 38844692
- [Result] Chinchilla M, Lulla A, Agans D, Chassman S, Gabrielian SE, Young AS. Pathways to social integration among homeless-experienced adults with serious mental illness: a qualitative perspective. BMC Health Serv Res. 2024 Oct 4;24(1):1180. doi: 10.1186/s12913-024-11678-6. PMID 39367388

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at the Greater Los Angeles VA 10/18/2021 - 6/24/2024.
Pre-assignment Details: Enrolled participants are provided with mobile monitoring. Mobile monitoring is the only group in this study.
Groups:
- mobile application: Participants use a mobile application on their smartphone that monitors and transmits mobile sensor and utilization data.
Period: Overall Study
Arm/Group | mobile application
Started | 87
Completed | 58
Not Completed | 29

BASELINE CHARACTERISTICS:
Arm/Group | Mobile Application
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 38
  White | 29
  More than one race | 3
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Passive Self-tracking of Mental Health
Description: Feasibility of passive self-tracking of mental health. The number of participants who completed the study.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | mobile application
Number analyzed (Participants) | 87
Participants | 58

2. Primary Outcome: Estimates of Sociability
Description: Use mobile sensor and phone utilization data to develop individualized estimates of sociability. There was an effort to calculate an estimate of sociability for each participant. Some participants had insufficient data collected to calculate an estimate. The intent is to determine the number of participants for whom this outcome can be estimated. The investigators report here on the number of participants for whom an estimate of sociability could be successfully calculated.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | mobile application
Number analyzed (Participants) | 87
Participants | 73

3. Primary Outcome: Identify Exacerbations of Psychiatric Symptoms
Description: Study the predictive value of using data on sociability, activities, and sleep to identify exacerbations of psychiatric symptoms. There was an effort to calculate identify exacerbations of psychiatric symptoms for each participant. Some participants had insufficient data collected to identify exacerbations. The intent is to determine the number of participants for whom this outcome can be estimated. The investigators report here on the number of participants for whom exacerbations of psychiatric symptoms could be successfully calculated.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | mobile application
Number analyzed (Participants) | 87
Participants | 85

4. Primary Outcome: Acceptability of Passive Self-tracking of Mental Health
Description: Acceptability of passive self-tracking of mental health. The number of participants who completed the study.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | mobile application
Number analyzed (Participants) | 87
Participants | 58

5. Primary Outcome: Safety of Passive Self-tracking of Mental Health
Description: Safety of passive self-tracking of mental health. The number of participants with a serious adverse event.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | mobile application
Number analyzed (Participants) | 87
Participants | 0

6. Primary Outcome: Estimates of Activities
Description: Use mobile sensor and phone utilization data to develop individualized estimates of activities. There was an effort to calculate an estimate of activity for each participant. Some participants had insufficient data collected to calculate an estimate. The intent is to determine the number of participants for whom this outcome can be estimated. The investigators report on the number of participants for whom an estimate of activity could be successfully calculated.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | mobile application
Number analyzed (Participants) | 87
Participants | 85

7. Primary Outcome: Estimates of Sleep
Description: Use mobile sensor and phone utilization data to develop individualized estimates of sleep. There was an effort to calculate an estimate of sleep for each participant. Some participants had insufficient data collected to calculate an estimate. The intent is to determine the number of participants for whom this outcome can be estimated. The investigators report here on the number of participants for whom an estimate of sleep could be successfully calculated.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | mobile application
Number analyzed (Participants) | 87
Participants | 85

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during participant enrollment. The enrollment period for participants was 9 months.
Description: Adverse events were monitoring in all participants.
Arm/Group | mobile application
All-Cause Mortality (participants affected / at risk) | 1/87
Serious Adverse Events (participants affected / at risk) | 0/87
Other Adverse Events (participants affected / at risk) | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT05023252/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT05023252/ICF_000.pdf